CLINICAL TRIAL: NCT01011920
Title: Randomized Phase II Trial On Primary Chemotherapy With High-Dose Methotrexate And High-Dose Cytarabine With Or Without Thiotepa, And With Or Without Rituximab, Followed By Brain Irradiation Vs. High-Dose Chemotherapy Supported By Autologous Stem Cells Transplantation For Immunocompetent Patients With Newly Diagnosed Primary CNS Lymphoma
Brief Title: Trial for Patients With Newly Diagnosed Primary Central Nervous System (CNS) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG32
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2016-07

CONDITIONS: Central Nervous System Lymphoma
Keywords: newly diagnosed primary central nervous system lymphoma
MeSH Terms: interventions — Methotrexate; Cytarabine; Rituximab; Thiotepa; Radiotherapy; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MTX+ AraC (Experimental): Arm A Methotrexate 3.5 g/m2 (0.5 g/m2 in 15 min. + 3 g/m2 in 3-hr infusion) d 1 Cytarabine 2 g/m2 1 hr infusion, twice a day (every 12 hs.) d 2 - 3
  Interventions: Drug: Methotrexate; Drug: Ara-C
- Ara-C +Rituximab (Experimental): Arm B Rituximab 375 mg/m2 conventional infusion d -5 & 0 Methotrexate 3.5 g/m2 0.5 g/m2 in 15 min. + 3 g/m2 in 3-hr infusion d 1 Cytarabine 2 g/m2 1 hr infusion, twice a day (every 12 hs.) d 2 - 3
  Interventions: Drug: Ara-C; Drug: Rituximab
- Ara-C + rituximab+thiotepa (Experimental): Arm C Rituximab 375 mg/m2 conventional infusion d -5 & 0 Methotrexate 3.5 g/m2 0.5 g/m2 in 15 min. + 3 g/m2 in 3-hr infusion d 1 Cytarabine 2 g/m2 1 hr infusion, twice a day (every 12 hs.) d 2 - 3 Thiotepa 30 mg/m2 30 min. Infusion d 4
  Interventions: Drug: Ara-C; Drug: Rituximab; Drug: Thiotepa
- WBRT 36 Gy +/- boost 9 Gy (Experimental): ARM D: WBRT with 36 Gy in the case of CR to primary chemotherapy or the same WBRT dose followed by a tumor-bed boost of 9 Gy with 1-2 cm of margin surrounding enhanced residual lesion (total tumor-bed dose 45 Gy) in patients who achieved a PR or SD after primary chemotherapy. Photons of 4-10 Mev, 180 cGy per day, 5 weekly fractions.
  Interventions: Radiation: radiotherapy
- BCNU + Thiotepa + APBSCT (Experimental): Arm E BCNU 400 mg/m2 in 500 ml saline sol 1-hr inf. day -6 Thiotepa 5 mg/kg in 250 ml saline sol 2-hr inf. every 12 hrs days -5 & -4 Reinfusion of PBSC ≥5 x 106 CD34+ cells/kg day 0
  Interventions: Drug: Thiotepa; Drug: BCNU; Other: APBSCT

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 3.5 g/m2 (0.5 g/m2 in 15 min. + 3 g/m2 in 3-hr infusion) on day 1, every 3 weeks for a maximum of 4 courses.
  Arms: MTX+ AraC
Drug: Ara-C — Cytarabine 2 g/m2 (1 hr infusion, twice a day every 12 hours), on d 2 - 3 every 3 weeks for a maximum of 4 courses
  Other Names: Cytarabine
  Arms: Ara-C + rituximab+thiotepa; Ara-C +Rituximab; MTX+ AraC
Drug: Rituximab — Rituximab 375 mg/m2 conventional infusion on day - 5 & 0 every 3 weeks for a maximum of 4 cycles
  Other Names: MabThera
  Arms: Ara-C + rituximab+thiotepa; Ara-C +Rituximab
Drug: Thiotepa — ARM C: Thiotepa 30 mg/m2 (30 min. Infusion) on day 4 every 3 weeks for a maximum of 4 courses ARM E: Thiotepa 5 mg/kg in 250 ml saline sol 2-hr inf. every 12 hrs days -5 & -4
  Arms: Ara-C + rituximab+thiotepa; BCNU + Thiotepa + APBSCT
Radiation: radiotherapy — Photons of 4-10 Mev, 180 cGy per day, 5 weekly fractions. Whole-brain will be irradiated by two opposite lateral fields including the first two cervical vertebras and the posterior two thirds of the orbits, which must be shielded after 30 Gy (after 36 Gy in the case of evident intraocular disease at diagnosis). Tumor-bed (boost or partial-brain RT) will be irradiated by 2 to 4 isocentric treatment fields based on tumor location, with all portals treated per each RT session.
  Arms: WBRT 36 Gy +/- boost 9 Gy
Drug: BCNU — BCNU 400 mg/m2 in 500 ml saline sol 1-hr inf. day -6
  Other Names: Carmustine
  Arms: BCNU + Thiotepa + APBSCT
Other: APBSCT — Autologous peripheral blood stem cell transplant (APBSCT)
  Arms: BCNU + Thiotepa + APBSCT

SUMMARY:
This is a multicenter open label randomized phase II trial.

Enrolled Primary Central Nervous System Lymphoma (PCNSL) patients will be stratified according to the IELSG score and randomized to receive one of the follows as primary chemotherapy:

* Arm A: Methotrexate (MTX) + Cytarabine (Ara-C)
* Arm B: MTX + Ara-C + rituximab
* Arm C: MTX + Ara-C + rituximab + thiotepa.

Chemotherapy will be administered every three weeks. The maximum number of chemotherapy induction courses will be 4. Patients in Stable Disease (SD) or better after two courses will receive two more courses of the same primary chemotherapy regimen. Stem-cells harvest will be performed in the three arms after the second course. After 4 courses response assessment will be performed.

Patients who will not achieve SD or better after the 4th course, as well as those who will experience Progressive Disease (PD) at any time and those who will not achieve a sufficient stem cell harvest, will receive Whole Brain Radiation Therapy (WBRT) 36-40 Gy +/- tumor bed boost of 9 Gy.

Patients who will achieve SD or better after the 4th course will be stratified according to objective response to primary chemotherapy and to primary chemotherapy regimen and randomly allocated to receive as consolidation therapy one of the follows:

* Arm D: WBRT 36 Gy +/- boost 9 Gy
* Arm E: Carmustine (BCNU) + Thiotepa + Autologous Peripheral Blood Stem Cell Transplant (APBSCT) Patients in Complete Response (CR) after WBRT or APBSCT will remain in follow-up. Patients who will not achieve a CR after WBRT will be managed according to physician's preferences. Patients who will not achieve a CR after APBSCT will be referred to WBRT.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological assessed diagnosis of non-Hodgkin's lymphoma.
* Diagnostic sample obtained by stereotactic or surgical biopsy, Cerebrospinal Fluid (CSF) cytology examination or vitrectomy.
* Disease exclusively localized into the central nervous system, CSF, cranial nerves or eyes.
* At least one measurable lesion.
* Previously untreated patients (previous or ongoing steroid therapy admitted).
* Age 18-65 years (with ECOG Performance Status 0-3) or 66-70 (with ECOG Performance Status 0-2).
* Adequate bone marrow, renal, cardiac, and hepatic function.
* Sexually active patients of childbearing potential agreeing in implementing adequate contraceptive measures during study participation.
* Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Patient-signed informed consent obtained before registration.

Exclusion Criteria:

* Patients with lymphomatous lesions outside the CNS.
* Patients with a previous non-Hodgkin lymphoma at any time.
* Previous or concurrent malignancies with the exception of surgically cured carcinoma in-situ of the cervix, carcinoma of the skin or other cancers without evidence of disease at least from 5 years.
* HBsAg and HCV positivity.
* HIV infection, previous organ transplantation or other clinically evident form of immunodeficiency.
* Concurrent treatment with other experimental drugs.
* Concurrent Pregnancy or lactation.
* Patients not agreeing to take adequate contraceptive measures during the study.
* Symptomatic coronary artery disease, cardiac arrhythmias uncontrolled with medication or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-11; Primary Completion 2015-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
response rate after primary chemotherapy and 2 years failure free survival at second randomization | 3 months, 2 years

SECONDARY OUTCOMES:
safety, as acute and long-term toxicity | Throughout all the active treatment period
overall survival | From entry onto trial until death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — San Raffaele H Scientific Institute, Milan, Italy; Gerald Illerhaus, MD, Study Chair — University Medical Center, Freiburg, Germany; Emanuele Zucca, MD, Principal Investigator — IOSI, Bellinzona, Switzerland
Locations (23):
- Germany (9):
  - University Hospital, Aachen
  - Universitätsklinikum Erlangen, Erlangen
  - "Klinik für Hämatologie Universitätsklinikum Essen", Essen
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Universitätskrankenhaus Hamburg-Eppendorf, Hamburg
  - Friedrich Schiller Universitaet Jena, Jena
  - Johannes Gutenberg Universität Mainz, Mainz
  - Technische Universität in München, München
  - Universitätsklinikum Ulm, Ulm
- Italy (11):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Spedali Civili, Brescia
  - San Raffaele H Scientific Institute, Milan
  - Ospedale Umberto I, Nocera Inferiore
  - Ospedale Civile S.Spirito, Pescara
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Nazionale dei Tumori Regina Elena, Roma
  - Università degli Studi La Sapienza, Roma
  - Humanitas, Rozzano
  - Ospedale Maggiore S. Giovanni Battista, Torino
  - Policlinico G.B. Rossi, Verona
- IOSI - Oncology Institute of Southern Switzerland, Bellinzona, Switzerland
- United Kingdom (2):
  - Nottingham City Hospital, Nottingham
  - Queen's Hospital, Romford

REFERENCES:
- [Derived] Ferreri AJM, Cwynarski K, Pulczynski E, Fox CP, Schorb E, La Rosee P, Binder M, Fabbri A, Torri V, Minacapelli E, Falautano M, Ilariucci F, Ambrosetti A, Roth A, Hemmaway C, Johnson P, Linton KM, Pukrop T, Sonderskov Gorlov J, Balzarotti M, Hess G, Keller U, Stilgenbauer S, Panse J, Tucci A, Orsucci L, Pisani F, Levis A, Krause SW, Schmoll HJ, Hertenstein B, Rummel M, Smith J, Pfreundschuh M, Cabras G, Angrilli F, Ponzoni M, Deckert M, Politi LS, Finke J, Reni M, Cavalli F, Zucca E, Illerhaus G; International Extranodal Lymphoma Study Group (IELSG). Whole-brain radiotherapy or autologous stem-cell transplantation as consolidation strategies after high-dose methotrexate-based chemoimmunotherapy in patients with primary CNS lymphoma: results of the second randomisation of the International Extranodal Lymphoma Study Group-32 phase 2 trial. Lancet Haematol. 2017 Nov;4(11):e510-e523. doi: 10.1016/S2352-3026(17)30174-6. Epub 2017 Oct 17. PMID 29054815
- [Derived] Ferreri AJ, Cwynarski K, Pulczynski E, Ponzoni M, Deckert M, Politi LS, Torri V, Fox CP, Rosee PL, Schorb E, Ambrosetti A, Roth A, Hemmaway C, Ferrari A, Linton KM, Ruda R, Binder M, Pukrop T, Balzarotti M, Fabbri A, Johnson P, Gorlov JS, Hess G, Panse J, Pisani F, Tucci A, Stilgenbauer S, Hertenstein B, Keller U, Krause SW, Levis A, Schmoll HJ, Cavalli F, Finke J, Reni M, Zucca E, Illerhaus G; International Extranodal Lymphoma Study Group (IELSG). Chemoimmunotherapy with methotrexate, cytarabine, thiotepa, and rituximab (MATRix regimen) in patients with primary CNS lymphoma: results of the first randomisation of the International Extranodal Lymphoma Study Group-32 (IELSG32) phase 2 trial. Lancet Haematol. 2016 May;3(5):e217-27. doi: 10.1016/S2352-3026(16)00036-3. Epub 2016 Apr 6. PMID 27132696